CLINICAL TRIAL: NCT07322471
Title: Efficacy and Safety of Flexible Ureteroscopy Versus Percutaneous Nephrolithotomy in Management of Staghorn Stones: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Flexible Ureteroscopy Versus Percutaneous Nephrolithotomy in Management of Staghorn Stones
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ammar Fathi Mohamed AlOrabi, Principle investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCNL vs FURS in staghorn stone
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Renal Stones
Keywords: PCNL; RIRS; staghorn stone; renal stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCNL group (Active Comparator): patients of this group will undergo percutanous nephrolithotomy
  Interventions: Procedure: Percutaneous nephrolithotomy
- FURS group (Active Comparator): Patients of this group will undergo flexible ureteroscopy
  Interventions: Procedure: Flexible ureteroscopy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — This intervention includes percutaneous nephrolithotomy for lithotripsy of staghorn stone
  Arms: PCNL group
Procedure: Flexible ureteroscopy — This intervention includes Flexible ureteroscopy for lithotripsy of staghorn stone
  Arms: FURS group

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is considered the treatment of choice for management of large renal calculi larger than 2 cm based on the yearly updated European Association of Urology (EAU) guidelines. However, PCNL is a challenging procedure which may be associated with several complications ranging from mild complications, such as urinary extravasation, leakage, infection and bleeding requiring transfusion to sever complications, such as sepsis, injury to surrounding organs, persistent hematuria and renal function impairment. The overall complication rate varies based on patient factors and surgical expertise.

Not only serious complications that defer some endourologists from performing PCNL but also such procedure is contraindicated and avoided by surgeons in cases of retrorenal colon, morbidly obese patients, spinal abnormalities and bleeding diathesis. Therefore, retrograde intrarenal surgery (RIRS) or flexible ureteroscopy (FURS) is increasingly recognized as an effective alternative, particularly for patients seeking a minimally invasive approach with a lower risk of complications.

The best practice in dealing with renal stones using FURS can be achieved via preoperative stenting for 2-4 weeks, negative urine culture, ureteral access sheath (UAS) usage and optimizing laser settings. Compared to PCNL, FURS is a less challenging procedure with low learning curve, less invasive and less bleeding. However, the high cost, including laser usage cost, presenting costs and multisession costs, in addition to the high risk of postoperative infection are considered as major drawbacks of FURS.

RIRS is emerging as an effective, safe, minimally invasive alternative to PCNL. Yet, the success of RIRS in comparison to PCNL, especially in a single session, is still questionable and there is no consensus about it.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Diagnosis of complete staghorn renal stones confirmed by non-contrast CT.
* Negative urine culture.

Exclusion Criteria:

* Congenital renal anomalies (e.g., horseshoe kidney, malrotation).
* Coagulopathy or uncorrected bleeding disorder.
* Pregnancy.
* Previous ipsilateral renal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 1 Month
  Stone-free rate (SFR), defined as no clinically significant residual stones on non-contrast 3-mm-cuts CT, measured as yes or no.

SECONDARY OUTCOMES:
Operative time | During the surgery
  Operative time is defined as time between starting the procedure and termination of it measured in minutes
Complications | 1 month
  Intra and postoperative complications, defined as complications happens intraoperative and postoperatively, graded by modified clavien-dindo classification
Radiation time | During the surgery
  Radiation time, defined as time in which ionizing radiation used intraoperatively, measured in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shebin El-Kom, Menoufia, Egypt